CLINICAL TRIAL: NCT03613077
Title: A Non-Interventional Study to Document the Use of Straumann BLX Implants in Daily Dental Practice
Acronym: BLX_NIS
Status: Completed | Type: Observational
Sponsor: Institut Straumann AG (Industry)
Responsible Party: Sponsor
Other Study IDs: CR2017-03
Record Dates: First submitted 2018-07-11; First posted 2018-08-02 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Surgical Operation With Implant of Artificial Internal Device
Keywords: Survival rate; Success rate; Straumann® BLX Implant Roxolid® SLActive®,

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: surgical placement of an endosteal implant — Subjects, male or female at least 18 years old, with the need of dental implant therapy and restoration according to the cleared indications for the implant

SUMMARY:
Prospective, multi-center, non-interventional observation to document the success and survival rates of Straumann BLX Implants used for tooth replacement in cleared indications up to 1 year after implant placement

DETAILED DESCRIPTION:
Objective of the study is to confirm the safety and performance of Straumann BLX Implants used for tooth replacement in cleared indications up to 12 months after implant placement. Implants used are Straumann® BLX Implant Roxolid® SLActive®. Regular Base (3.5 mm): implant diameters 3.75 and 4.5mm, in lengths 6, 8, 10, 12,14, 16 and 18 mm Wide Base (4.5 mm): diameter 5.5 mm in lengths 6, 8, 10 and 12 mm

ELIGIBILITY:
Inclusion Criteria:

* Patients seeking an implant supported restoration
* all patients with conditions that are in accordance with the IFU
* Patients must provide their informed consent for study participation and must be willing and able to attend control visits
* Patients need to be at least 18 years old

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients seeking an implant supported restoration
Sampling Method: Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2018-05-14 (Actual); Primary Completion 2020-02-02 (Actual); Study Completion 2025-08-21 (Actual)

PRIMARY OUTCOMES:
Implant success rate at one year post implant placement | 12 months follow-up period after implantation
  Measured in percent
Implant survival rate at one year post implant placement | 12 months follow-up period after implantation
  Measured in percent

SECONDARY OUTCOMES:
Prosthetic success at 12 months post implant placement | 12 months follow-up period after implantation
  Measured in percent
Prosthetic survival at 12 months post implant placement | 12 months follow-up period after implantation
  Measured in percent

CONTACTS AND LOCATIONS:
Overall Officials: Christian Walter, Prof. Dr.Dr., Principal Investigator — Mediplus Praxisklinik
Locations (1):
- Mediplus Praxisklinik, Mainz, Germany

IPD SHARING:
Plan to Share IPD: No